CLINICAL TRIAL: NCT02833298
Title: Post Sustained Virological Response (SVR) Hepatocellular Carcinoma (HCC) Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 16-1542
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma; HCC; Hepatitis C; HCV
Keywords: Sustained Virological Response; SVR; patient navigation; screening; HCC; HCV
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Automated reminders (Experimental): Patient will be contacted for automated reminders within one month before the six-month interval indicating they are due for HCC screening.
  Interventions: Behavioral: Automated reminders
- Patient navigation (Experimental): The patient navigator will coordinate with the provider and subject to schedule the appropriate office visit and imaging for HCC screening as needed within one month before the test is due.
  Interventions: Behavioral: Patient navigation

INTERVENTIONS:
Behavioral: Automated reminders — At the time consent is obtained, members of the research team will collect data about how a subject prefers to be contacted for automated reminders (i.e. text messages, postcard, email, MyChart)
  Arms: Automated reminders
Behavioral: Patient navigation — The patient navigator will attempt to provide a reminder to the subject one to three days before the scheduled imaging and also offer to accompany the subject to the test.
  Arms: Patient navigation

SUMMARY:
Approximately half of the patients receiving treatment for chronic hepatitis C virus (HCV) infection in the United States have advanced liver disease. Patients with advanced fibrosis/cirrhosis who achieve a sustained virological response (SVR) to treatment and are clinically cured of HCV continue to have an elevated risk of developing hepatocellular carcinoma (HCC). According to guidelines from several professional societies and from the American Association for the Study of Liver Diseases (AASLD), in particular, patients with advanced fibrosis/cirrhosis should undergo life-long bi-annual screening for incident HCC whether they achieve an SVR, or not. The number of patients who need post-SVR HCC screening has risen dramatically in recent years due to the confluence of three factors: Increased screening for HCV, which has allowed more people to realize that they have this often "silent" infection; the availability of safe and highly effective direct acting antiviral drugs (DAAs) for HCV, which has allowed a much higher percentage of treated patients to achieve an SVR; and the long duration of HCV infection in many patients, which has allowed enough time for advanced fibrosis/cirrhosis to develop. To investigate post-SVR patients in the era of DAAs and to promote HCC screening, the objective of this study is to conduct a randomized, unblinded, two-arm prospective intervention trial comparing rates of HCC screening between patients randomized to either personalized patient navigation or automated reminders (e.g. electronic or mailed). Both interventions represent improved care over current standard of care (no patient navigation or automated reminders). There is no evidence to suggest one intervention is better than the other. Healthcare providers who agree to participate in the study will be contacted to confirm the liver disease status of their patients and during the clinical trial the providers of patients in both arms of the trial will be sent reminders about the need to schedule patients for screening visits.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years old
* history of HCV infection treated in 2011 or after with direct acting antiviral therapy
* achieved ≥SVR-12 as defined as no detectable virus 12 weeks or longer after the cessation of therapy
* FIB-4 ≥3.25
* no history of HCC prior to treatment
* HCV provider deems a subject eligible for HCC surveillance according to AASLD criteria
* able to understand and speak English
* willing to sign the informed consent
* have a working phone number or e-mail to reach them
* no history of liver transplantation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
HCC screening rates | every 6 months until death - average of 5 years
  Ratio of Number of on-time screening visits to number of missed screening visits

SECONDARY OUTCOMES:
Adherence to HCC Surveillance | every 6 months until death - average of 5 years
  Percentage for patients completing timely screening visit
Rates of HCC | every 6 months until death - average of 5 years
  New incidences of HCC
Incidence of Death | every 6 months until death - average of 5 years
  Incidence of death
Incidence of liver transplant | every 6 months until death - average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ponni Perumalswami, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No